CLINICAL TRIAL: NCT00556062
Title: The Clinical Trial for Three Consecutive Lots of Influenza Split Vaccine Anflu by Randomized, Double-Blind and Controlled Design
Brief Title: Phase IV Clinical Trial of an Influenza Split Vaccine Anflu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-INF-4005
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- 1: Lot 1 (Experimental)
  Interventions: Biological: seasonal split influenza vaccine
- 2: Lot 2 (Experimental)
  Interventions: Biological: seasonal split influenza vaccine
- 3: Lot 3 (Experimental)
  Interventions: Biological: seasonal split influenza vaccine
- 4: control vaccine (Active Comparator)
  Interventions: Biological: seasonal split influenza vaccine

INTERVENTIONS:
Biological: seasonal split influenza vaccine — 0.5 ml/dose, containing 45 μg influenza HA antigens, 15 μg each subtype; one dose regime
  Arms: 1: Lot 1
Biological: seasonal split influenza vaccine — 0.5 ml/dose, containing 45 μg influenza HA antigens, 15 μg each subtype; one dose regime
  Arms: 2: Lot 2
Biological: seasonal split influenza vaccine — 0.5 ml/dose, containing 45 μg influenza HA antigens, 15 μg each subtype; one dose regime
  Arms: 3: Lot 3
Biological: seasonal split influenza vaccine — 0.5 ml/dose, containing 45 μg influenza HA antigens, 15 μg each subtype; one dose regime
  Arms: 4: control vaccine

SUMMARY:
To evaluate the safety and immunogenicity of the three consecutive lots of an seasonal split influenza vaccine Anflu in adults, a randomized, double-blind and controlled clinical trial was conducted in 560 subjects in Tianjin City of China.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-60 years old
* Be able to show legal identity card for the sake of recruitment Without vaccination history of seasonal split influenza vaccine in the recent 3 years
* Not participate in any other clinical trials during the study
* Not receive any immunosuppressive agents during and one month prior to the study
* Be able to understand and sign the informed consent.

Exclusion Criteria:

* Woman： Who breast-feeding or planning to become pregnant during the study
* Any history of allergic reactions; was allergic to any component of the vaccine, such as eggs or ovalbumin
* Any history of severe adverse reactions to vaccines, such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Autoimmune disease or immunodeficiency
* Acute episode of chronic diseases or conditions, including chronic hepatitis, hypertension, diabetes mellitus and cardiovascular diseases
* Guillain-Barre Syndrome
* Women subjects with positive urinary pregnancy test
* Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
* Axillary temperature >37.0 centigrade at the time of dosing
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 566 (Actual)
Dates: Start 2007-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Haemagglutination-inhibition (HI) antibody titer of influenza A H1N1, influenza A H3N2 and influenza B | 0, 21 days

SECONDARY OUTCOMES:
local and systematic adverse reactions after vaccination | within 3 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Zhilun Zhang, Principal Investigator — Tianjin centers for Disease Control and Prevention